CLINICAL TRIAL: NCT01464424
Title: Assessment of Late Day IOP Control in Subjects With Open-Angle Glaucoma or Ocular Hypertension Treated With Travoprost 0.004% (TRAVATAN® Z) or Bimatoprost 0.01% (LUMIGAN®)
Brief Title: Assessment of Intraocular Pressure (IOP) Control in Subjects With Open-Angle Glaucoma or Ocular Hypertension Treated With Travoprost 0.004% (TRAVATAN® Z) or Bimatoprost 0.01% (LUMIGAN®)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RDG-10-003
Record Dates: First submitted 2011-11-01; First posted 2011-11-03 (Estimated); Results first posted 2013-09-04 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Glaucoma; Ocular Hypertension; Open-Angle Glaucoma
Keywords: Glaucoma; Ocular Hypertension; Open-Angle Glaucoma; Intraocular Pressure
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Glaucoma, Open-Angle | interventions — Travoprost; Ophthalmic Solutions; Bimatoprost

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TRAVATAN, then LUMIGAN (Other): Travoprost 0.004% ophthalmic solution (TRAVATAN), 1 drop to the study eye once daily every evening at 8:00 pm for 6 weeks, followed by bimatoprost 0.01% ophthalmic solution (LUMIGAN), same dose, same duration, as randomized, for a total duration of 12 weeks
  Interventions: Drug: Travoprost 0.004% ophthalmic solution; Drug: Bimatoprost 0.01% ophthalmic solution
- LUMIGAN, then TRAVATAN (Other): Bimatoprost 0.01% ophthalmic solution (LUMIGAN), 1 drop to the study eye once daily every evening at 8:00 pm for 6 weeks, followed by travoprost 0.004% ophthalmic solution (TRAVATAN), same dose, same duration, as randomized, for a total duration of 12 weeks
  Interventions: Drug: Travoprost 0.004% ophthalmic solution; Drug: Bimatoprost 0.01% ophthalmic solution

INTERVENTIONS:
Drug: Travoprost 0.004% ophthalmic solution
  Other Names: TRAVATAN® Z
Drug: Bimatoprost 0.01% ophthalmic solution
  Other Names: LUMIGAN®

SUMMARY:
The purpose of this study was to assess efficacy and tolerability of travoprost 0.004% vs. bimatoprost 0.01% during the after office hour period (4 pm to 8 pm) in subjects with open-angle glaucoma or ocular hypertension after 6 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of open-angle glaucoma (OAG) or ocular hypertension (OHT) in at least one eye.
* Non-study eye: Intraocular pressure (IOP) able to be controlled with no pharmacologic therapy or on the study medicine alone.
* Willing to discontinue the use of all other ocular hypotensive medications prior to receiving study medication and for the entire course of the study.
* Able to follow instructions, self instill study article, and attend all study visits.
* Best-corrected Snellen visual acuity of 20/200 or better in each eye.
* Sign Ethics Committee reviewed and approved informed consent form.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Known medical history of allergy, hypersensitivity or poor tolerance to any component of the preparations used in this study.
* Any abnormality preventing applanation tonometry in either eye.
* Dry eye previously or currently being treated with punctal plugs, punctal cautery, Restasis®, or topical ocular corticosteroids.
* Concurrent infectious/noninfectious conjunctivitis, keratitis or uveitis in either eye.
* Intraocular conventional or laser surgery >3 months prior to consent.
* Risk of visual field or visual acuity worsening as a consequence of participation in the study, in the investigator's best judgment.
* Progressive retinal or optic nerve disease from any cause.
* Use of any systemic medications known to affect IOP which have not been on a stable course for at least 7 days prior to Screening or an anticipated change in dosage during the course of the study.
* Any clinically significant, serious, or severe medical condition.
* Women of childbearing potential who are pregnant, lactating, or not using reliable means of birth control.
* Participation in any other study within 30 days prior to Screening.
* Use of any systemic (oral), injectable or topical steroids.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2011-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doug Hubatsch, MS, Study Director — Alcon Research

REFERENCES:
- [Derived] DuBiner HB, Hubatsch DA. Late-day intraocular pressure-lowering efficacy and tolerability of travoprost 0.004% versus bimatoprost 0.01% in patients with open-angle glaucoma or ocular hypertension: a randomized trial. BMC Ophthalmol. 2014 Nov 28;14:151. doi: 10.1186/1471-2415-14-151. PMID 25432143

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 2 study centers located in the US.
Pre-assignment Details: This reporting group includes all enrolled subjects. A washout-period based on prior medication preceded Period 1 dispense.
Period: Period 1, First 6 Weeks
Arm/Group | TRAVATAN, Then LUMIGAN | LUMIGAN, Then TRAVATAN
Started | 42 | 42
Completed | 42 | 41
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Period 2, Second 6 Weeks
Arm/Group | TRAVATAN, Then LUMIGAN | LUMIGAN, Then TRAVATAN
Started | 42 | 41
Completed | 42 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This reporting group includes all enrolled subjects.
Groups:
- Overall: Travoprost 0.004% and bimatoprost 0.01% in cross-over fashion, as randomized, 6 weeks each
Arm/Group | Overall
Number analyzed (Participants) | 84
Age Continuous [Mean (Standard Deviation); unit: years] | 58.7 (11.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 29
Region of Enrollment [Number; unit: participants]
  United States | 84

OUTCOME MEASURES:

1. Secondary Outcome: Mean IOP at Each After Office Hour Evaluation Timepoint
Description: IOP was measured at three after office hour evaluation time points (4 pm, 6 pm, and 8 pm). The three timepoints correspond to 20, 22, and 24 hours post dose. Efficacy analysis was performed for one eye only, i.e., the designated study eye.
Time Frame: Week 6: 4 pm, 6 pm, 8 pm
Population: Per protocol: All subjects who received study medication, completed all study visits as per the protocol timelines and criteria, and satisfied inclusion/exclusion criteria.
Measure: Mean (Standard Deviation); unit: millimeters mercury (mmHg)
Groups:
- TRAVATAN: Travoprost 0.004% ophthalmic solution, 1 drop to the study eye once daily every evening at 8:00 pm for 6 weeks
- LUMIGAN: Bimatoprost 0.01% ophthalmic solution, 1 drop to the study eye once daily every evening at 8:00 pm for 6 weeks
Arm/Group | TRAVATAN | LUMIGAN
Number analyzed (Participants) | 81 | 81
millimeters mercury (mmHg)
  4 pm (20 hours post dose) | 17.74 (3.099) | 17.08 (2.808)
  6 pm (22 hours post dose) | 17.52 (2.836) | 17.32 (3.055)
  8 pm (24 hours post dose) | 17.06 (2.840) | 17.26 (2.890)

2. Primary Outcome: Overall Mean Intraocular Pressure (IOP)
Description: IOP was measured at three after office hour evaluation time points (4 pm, 6 pm, and 8 pm) for an overall mean. The three timepoints correspond to 20, 22, and 24 hours post dose. Efficacy analysis was performed for one eye only, i.e., the designated study eye. Per-protocol dataset was pre-specified for this non-inferiority analysis.
Time Frame: Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters mercury (mmHg)
Arm/Group | TRAVATAN | LUMIGAN
Number analyzed (Participants) | 81 | 81
millimeters mercury (mmHg) | 17.45 (2.664) | 17.22 (2.605)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study.
Description: Adverse events were obtained as solicited comments from the study subjects and as observations by the Study Investigator as outlined in the study protocol. This reporting group includes all enrolled subjects.
Arm/Group | TRAVATAN | LUMIGAN
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/84
Other Adverse Events (participants affected / at risk) | 0/84 | 0/84

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.